CLINICAL TRIAL: NCT06712472
Title: Randomized Phase III Trial Testing Maintenance Olaparib Versus Observation After Adjuvant Chemoradiation for p53abn Endometrial Cancer
Acronym: RAINBO-RED
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-503886-44-00; 2023/3603 (Other: CSET number)
Record Dates: First submitted 2024-11-26; First posted 2024-12-02 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Endometrial Cancer; p53abn
MeSH Terms: conditions — Endometrial Neoplasms | interventions — olaparib; BID protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard arm (No Intervention)
- Experimental arm (Experimental)
  Interventions: Drug: Olaparib (300 mg BID)

INTERVENTIONS:
Drug: Olaparib (300 mg BID) — Olaparib 300mg Bid during one year.
  Arms: Experimental arm

SUMMARY:
The RAINBO program is a studies group which proposes personalized treatment of patients suffering from endometrial cancer according to their molecular profile.

the RAINBO-RED study allows observation or maintenance treatment with targeted therapy for one year (olaparib). This after standard therapy. The goal is to improve recurrence-free survival of patients treated with Olaparib.

ELIGIBILITY:
Key inclusion criteria for RAINBO program:

* Histologically confirmed diagnosis of EC (all grades and the following histologic subtypes : endometrioid, serous, clear cell, de-/undifferentiated carcinomas, and uterine carcinosarcoma).
* Molecular classification performed following the diagnostic algorithm described in WHO 2020 (adapted from Vermij et al.)
* TLH-BSO or TAH-BSO with or without lymphadenectomy or sentinel node biopsy, without macroscopic residual disease after surgery
* No distant metastases as determined by pre-surgical or post-surgical imaging (CT scan of chest, abdomen and pelvis or PET-CT scan)
* Written informed consent prior to any study specific procedures
* Age >= 18 years
* Patients must have a life expectancy ≥ 16 weeks
* Patients must be accessible for treatment and follow-up
* Written informed consent for one of the RAINBO trials and the overarching research project according to the local Ethics Committee requirements.

Inclusion criteria specific for p53abn-RED Trial:

* WHO Performance score 0-1
* Histologically confirmed Stage I to III EC with myometrial invasion
* Molecular classification: p53abn EC*
* Body weight > 30 kg
* Patient must receive or have received a sequential radiotherapy and chemotherapy preferably given according to the PORTEC-3 regimen and should be started within 6 to 8 weeks after surgery and no later than 10 weeks: two cycles of intravenous cisplatin 50mg/m² in the first and fourth week of the pelvic external beam radiotherapy (EBRT) +/- vaginal brachytherapy followed by four cycles of intravenous carboplatin AUC 5 and paclitaxel 175 mg/m² at 21-day intervals.

However the sequence of chemotherapy , number of cycles and inclusion of cisplatin may be altered according to local practice at the investigator's discretion.

This may include;

* 4 cycles carboplatin & paclitaxel before or after radiotherapy with 2 cycles cisplatin
* 4 cycles carboplatin & paclitaxel before or after radiotherapy (no cisplatin)
* 6 cycles carboplatin & paclitaxel before or after radiotherapy (no cisplatin)

  * Patients registered after their standard treatment must:
  * provide a tumor assessment performed within the 4 weeks before the start of RT/CT. This will be considered as the M0.
  * have started RT/CT 6 to 8 weeks after surgery. A maximum gap of 10 weeks is accepted.
  * be randomized within two weeks before maintenance or observation.
  * Adequate systemic organ function: Patients must have normal organ and bone marrow function measured within 28 days prior to administration of study treatment as defined below:

    * Creatinine clearance (> 50 cc/min): Patients must have creatinine less than 1.5 ULN or calculated creatinine clearance estimated of ≥ 51 mL/min using the Cockcroft-Gault equation or based on a 24 hour urine test. Estimated creatinine clearance = (140-age [years]) x weight (kg) (x F) / serum creatinine (mg/dL) x 72
    * Adequate bone marrow function : hemoglobin ≥10.0 g/dl with no blood transfusion in the past 28 days, Absolute neutrophil count (ANC) ≥1.5 x 109/l, platelet count ≥ 100 x 109/l.
    * Adequate liver function: bilirubin ≤1.5 x institutional upper limit of normal (ULN). This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
    * ALT (SGPT) and/or AST (SGOT) ≤2.5 x ULN
  * *Molecular classification must be performed according to the diagnostic algorithm presented in the WHO 2020 (Vermij et al. 2020). For the p53abn-RED trial this means that MMR and POLE status must be determined, and must be pMMR and POLE wildtype (or non-pathogenic) for inclusion. For details on the molecular classification see 7.1: Diagnostic algorithm for molecular classification.
  * Patient should understand, sign, and date the written informed consent form prior to any protocol-specific procedures performed. Patient should be able and willing to comply with study visits and procedures as per protocol.
  * Patients must be affiliated to a social security system or beneficiary of the same

Exclusion Criteria:

Exclusion criteria for RAINBO program

* FIGO Stage IV disease of any histology even if there is no evidence of disease after surgery
* Prior pelvic irradiation

Exclusion criteria specific for p53abn-RED Trial:

* Other malignancy unless curatively treated with no evidence of disease for ≥5 years except: adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS), Stage 1, grade 1 endometrial carcinoma.
* Resting ECG indicating uncontrolled, potentially reversible cardiac conditions, as judged by the investigator (eg., unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, QTcF prolongation >500 ms, electrolyte disturbances, etc.), or patients with congenital long QT syndrome.
* Persistent toxicities (>Common Terminology Criteria for Adverse Event (CTCAE) grade 2) caused by previous cancer therapy, excluding alopecia.
* Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV).
* Patients receiving any systemic chemotherapy or radiotherapy (except for palliative reasons) within 3 weeks prior to study treatment
* Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on High Resolution Computed Tomography (HRCT) scan or any psychiatric disorder that prohibits obtaining informed consent.
* Major surgical procedure (as defined by the Investigator) within 2 weeks prior randomization and patients must have recovered from any effects of any major surgery.
* Significant traumatic injury within 4 weeks of the first dose of olaparib.
* History of allogenic organ transplantation.
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
* Patient with severe hepatic impairment
* Any previous treatment with a PARP inhibitor, including olaparib.
* History of active primary immunodeficiency
* History or evidence of hemorrhagic disorders within 6 months prior to randomization
* Patients with myelodysplastic syndrome/acute myeloid leukemia history or with features suggestive of MDS/AML.
* Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT)
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immuno-deficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Concomitant use of known strong CYP3A inhibitors (eg. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (eg. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting olaparib is 2 weeks.
* Concomitant use of known strong (eg. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers (eg. bosentan, efavirenz, modafinil). The required washout period prior to starting olaparib is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
* Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
* Medical or psychological condition which in the opinion of the investigator would not permit the patient to complete the study or sign meaningful informed consent.
* Patient under guardianship or deprived of his liberty by a judicial or administrative decision or incapable of giving its consent
* Patients with a known hypersensitivity to olaparib or any of the excipients of the product.
* Treatment with an unlicensed or investigational product within 4 weeks of trial entry.
* Breastfeeding patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 554 (Estimated)
Dates: Start 2024-06-26 (Actual); Primary Completion 2030-06 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence-Free survival | 3 years
  To assess whether maintenance therapy with olaparib improves recurrence-free survival (RFS), as compared to observation after chemo-radiotherapy in patients with p53abn HREC

CONTACTS AND LOCATIONS:
Locations (15):
- France (15):
  - Centre Hospitalier D'Albi, Albi
  - Institut Cancerologie de L'Ouest-Angers, Angers
  - Chu Besancon, Besançon
  - Centre Hospitalier de Carcassonne, Carcassonne
  - Chu Dijon, Dijon
  - Groupe Hospitalier Mutualiste de Grenoble, Grenoble
  - CHU De LIMOGES, Limoges
  - Centre LEON BERARD, Lyon
  - Institut Paoli Calmettes, Marseille
  - Centre Antoine LACASSAGNE, Nice
  - Institut Marie-Curie, Paris
  - Hopital Cochin, Paris
  - INSTITUT CANCEROLOGIE DE L'OUEST-St HERBLAIN, Saint-Herblain
  - Clinique Sainte Anne, Strasbourg
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No